CLINICAL TRIAL: NCT00290719
Title: A Phase I/II Study to Evaluate Safety and Efficacy in Patients Who Have Resectable Esophageal Cancer and Are Treated With Neoadjuvant Cisplatin, Irinotecan (CPT-11) ZD1839 (IRESSA), and Radiotherapy Followed by Surgical Resection
Brief Title: Gefitinib, Cisplatin, Irinotecan, and Radiation Therapy Before Surgery in Treating Patients With Esophageal Cancer or Gastroesophageal Junction Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456200; UCSF-034510; ZENECA-1839US/0244
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Gefitinib; Irinotecan; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: gefitinib
Drug: irinotecan hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving gefitinib together with chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I/II trial is studying the side effects of gefitinib when given together with cisplatin, irinotecan, and radiation therapy before surgery and to see how well they work in treating patients with esophageal cancer or gastroesophageal junction cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the pathologic response (complete and partial) in patients with resectable esophageal or gastroesophageal junction cancer treated with neoadjuvant gefitinib, cisplatin, irinotecan hydrochloride, and radiotherapy followed by surgical resection.

Secondary

* Assess the safety and toxicity of this regimen in these patients.
* Evaluate objective tumor response in patients treated with this regimen.
* Determine the rate of complete resection in patients treated with this regimen.
* Determine surgical morbidity and mortality in patients treated with this regimen.

OUTLINE: This is an open-label study.

* Induction phase: Patients receive oral gefitinib once daily on days 1-14. Patients with stable or responding disease proceed to neoadjuvant chemoradiotherapy.
* Neoadjuvant chemoradiotherapy: Patients receive gefitinib as in the induction phase beginning in week 4 and continuing through the last day of radiotherapy. Patients also receive cisplatin IV over 1 hour and irinotecan hydrochloride IV over 30 minutes on days 22, 29, 43, and 50 and undergo radiotherapy once daily, 5 days a week, for 5 weeks (total of 25 doses).
* Surgery: Within 4-8 weeks after completion of neoadjuvant chemoradiotherapy, patients with stable or responding disease undergo an esophagectomy and lymph node dissection. Patients with a progressive or unresectable disease are removed from the study.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma (AC) or squamous cell carcinoma of the esophagus

  * AC of the gastroesophageal junction allowed
* Tumor must be considered surgically resectable (T1-3, NX)

  * No early-stage cancer (T1, N0)
* The following lymph node (LN) criteria are considered acceptable:

  * Regional thoracic LN metastases (N1)
  * LN metastases levels 15 to 20 measured as ≤ 1.5 cm by CT scan
  * Supraclavicular LN not palpable on clinical examination measured as ≤ 1.5 cm by CT scan
* No distant metastases (M0)

PATIENT CHARACTERISTICS:

* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Creatinine clearance ≥ 50 mL/min
* Creatinine serum level ≤ CTC grade 2
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST < 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No known severe hypersensitivity to gefitinib or any of its excipients
* No evidence (except asymptomatic chronic stable radiographic changes) of clinically active interstitial lung disease
* No pulmonary fibrosis, Gilbert's disease, uncontrolled diabetes mellitus, or unstable angina
* No New York Heart Association class III or IV heart disease
* No other concurrent malignancies or malignancies diagnosed within the past 5 years except basal cell carcinoma or carcinoma in situ of the cervix
* No serious active or uncontrolled infection, systemic disease, psychiatric illness, or other medical condition that would preclude study participation
* No evidence of any significant clinical disorder or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for esophageal cancer
* No prior radiotherapy that would overlap the study treatment fields
* Recovered from prior major surgery
* No nonapproved or investigational drugs within the past 30 days
* No concurrent phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital, or Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pathological response (complete and partial) post-operatively

SECONDARY OUTCOMES:
Safety and toxicity post-operatively
Response rate 2 weeks into treatment, pre-operatively, and post-operatively
Completeness of resection post-operatively
Surgical morbidity and mortality post-operatively
Compare the effects of gefitinib on biomarkers that effect EGF signaling and genomic composition of tumor samples before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States